CLINICAL TRIAL: NCT01996735
Title: The Effect of Ticagrelor on the Adenosine System
Brief Title: Ticagrelor and Adenosine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NL43379.091.13
Record Dates: First submitted 2013-04-26; First posted 2013-11-27 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2013-02

CONDITIONS: Healthy
Keywords: Endothelial function; Adenosine receptor stimulation
MeSH Terms: interventions — Ticagrelor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ticagrelor 180 mg single dose (Active Comparator): Ticagrelor 180 mg single dose
  Interventions: Drug: Ticagrelor 180 mg single dose
- Placebo (Placebo Comparator): Placebo single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ticagrelor 180 mg single dose
  Arms: Ticagrelor 180 mg single dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
Preclinical studies have shown that the P2Y12 receptor antagonist ticagrelor can increase the extracellular concentration of the endogenous nucleoside adenosine by inhibiting the cellular uptake of adenosine via the equilibrative nucleoside transporter (ENT). This mechanism can contribute to the beneficial effects and to the side effects (dyspnea) of ticagrelor in patients with an acute myocardial infarction. In the current research proposal, we aim to investigate whether ticagrelor increases adenosine receptor stimulation in humans in vivo by ENT inhibition.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* Age 18-40 years
* Healthy
* Written informed consent

Exclusion Criteria:

* Smoking
* Hypertension (Blood pressure >140 mmHg and/or >90 mmHg - SBP/DBP-)
* Diabetes Mellitus (fasting glucose > 7.0 mmol/L or random > 11.0 mmol/L)
* History of any cardiovascular disease
* History of chronic obstructive pulmonary disease (COPD) or asthma
* Bleeding tendency
* Concomitant use of medication
* Renal dysfunction (MDRD < 60 ml/min)
* Liver enzyme abnormalities (ALAT > twice upper limit of normality)
* Thrombocytopenia (<150*109/ml)
* Second/third degree AV-block on electrocardiography

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2013-04; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Forearm blood flow response | 2 hours after intake of ticagrelor/placebo
  Forearm blood flow response to the intrabrachial administration of incremental dosages of adenosine, after treatment with ticagrelor compared to placebo. The forearm blood flow will be measured by plethysmography.
Forearm blood flow response | Directly after 2 and 5 minutes of forearm ischemia
  Directly after 2 and 5 minutes of forearm ischemia.The forearm blood flow will be measured by plethysmography.

SECONDARY OUTCOMES:
Forearm blood flow respons | Directly after administration of dipyridamole
  Forearm blood flow response to the intrabrachial administration of incremental dosages of dipyridamole, after treatment with ticagrelor compared to placebo. The forearm blood flow will be measured by plethysmography
ex-vivo adenosine uptake in isolated erythrocytes | 2 hours after intake of studymedication
  To study whether ticagrelor inhibits the ex-vivo adenosine uptake in isolated erythrocytes

CONTACTS AND LOCATIONS:
Overall Officials: N. Riksen, MD, PhD, Principal Investigator — Radboud University Medical Center; G. Rongen, MD, PhD, Principal Investigator — Radboud University Medical Center; M. Gomes, MD, PhD, Principal Investigator — Dept Cardiology, Canisius Wilhelmina Hospital Nijmegen; S. El Messaoudi, MD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] van den Berg TN, El Messaoudi S, Rongen GA, van den Broek PH, Bilos A, Donders AR, Gomes ME, Riksen NP. Ticagrelor Does Not Inhibit Adenosine Transport at Relevant Concentrations: A Randomized Cross-Over Study in Healthy Subjects In Vivo. PLoS One. 2015 Oct 28;10(10):e0137560. doi: 10.1371/journal.pone.0137560. eCollection 2015. PMID 26509673